CLINICAL TRIAL: NCT00528398
Title: Phase II Trial Utilizing Idarubicin in Combination With High Dose Ara-C for Induction Therapy for Adult Acute Myelogenous Leukemia (AML)
Brief Title: Idarubicin and High-Dose Cytarabine in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 93139; P30CA033572 (NIH); CHNMC-93139; CHNMC-93139-94-03-1; CDR0000564537 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Leukemia
Keywords: adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Congenital Abnormalities | interventions — Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (idarubicin, cytarabine) (Experimental): Patients receive cytarabine IV over 3 hours every 12 hours on days 1-4 and idarubicin IV over 5-10 minutes on days 1-3. Patients undergo bone marrow aspirate and biopsy 7 days after completion of induction chemotherapy. Patients with > 25% cellular biopsy or > 10% abnormal cells on aspirate receive 4 more doses of cytarabine and 1 dose of idarubicin.
  Interventions: Drug: cytarabine; Drug: idarubicin

INTERVENTIONS:
Drug: cytarabine
  Other Names: Cytosine Arabinoside; Cytosar-U; Depocyt
Drug: idarubicin
  Other Names: 4-demethoxydaunorubicin; Idamycin; Zavedos

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving idarubicin together with high-dose cytarabine works in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete remission rate (CR).
* Determine the proportion of patients who are bone marrow-positive at day 7 post-induction chemotherapy.
* Further evaluate the toxicity of this regimen.

OUTLINE: Patients receive cytarabine IV over 3 hours every 12 hours on days 1-4 and idarubicin IV over 5-10 minutes on days 1-3. Patients undergo bone marrow aspirate and biopsy 7 days after completion of induction chemotherapy. Patients with > 25% cellular biopsy or > 10% abnormal cells on aspirate receive 4 more doses of cytarabine and 1 dose of idarubicin.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Newly diagnosed acute myeloid leukemia (AML)

  * Morphologic proof (bone marrow aspirate smears or touch prep of marrow biopsy) of disease
  * FAB M0, M1, M2, M4, M5a, M5b, M6a, M6b, and M7 disease
* Previously untreated with radiotherapy or chemotherapy

  * Patients with treatment-related leukemia are eligible even if they have received prior chemotherapy and radiotherapy
* Patients with prior myelodysplastic syndrome are eligible
* Extramedullary leukemia allowed
* AML with lymphoid markers allowed

Exclusion criteria:

* Blastic transformation of chronic myelogenous leukemia
* Biphenotypic leukemia
* FAB M3 disease (acute promyelocytic leukemia)

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 weeks
* Total bilirubin < 1.5 g/dL
* AST and ALT < 5 times upper limit of normal (ULN)
* Creatinine < 1.5 mg/dL OR creatinine clearance > 70 mL/min
* Ejection fraction ≥ 50% by MUGA unless decreased ejection fraction is secondary to leukemia infiltration
* HIV antibody-negative

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* Prior hydroxyurea or corticosteroids allowed
* At least 48 hours since prior and no concurrent itraconazole or fluconazole

Exclusion criteria:

* More than 300 mg/m² of prior daunorubicin or equivalent dose of anthracycline

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 1994-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S. Stein, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Idarubicin, Cytarabine): All patients were analyzed together.
Period: Overall Study
Arm/Group | Treatment (Idarubicin, Cytarabine)
Started | 111
Completed | 111
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Idarubicin, Cytarabine)
Number analyzed (Participants) | 111
Age, Continuous [Median (Full Range); unit: years] | 43 [17 to 60]
Gender [Count of Participants; unit: Participants]
  Female | 50
  Male | 61
Diagnosis [Count of Participants; unit: Participants]
  De Novo AML | 80
  AML Secondary to Chemotherapy | 6
  AML Evolved from MDS | 25

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR)
Description: The peripheral blood neutrophil count is >= 1.5 x 10^9 / L and platelets more than 100 x 10^9 / L. Leukemia blast cells are not present in the peripheral blood. The cellularity of the bone marrow is more than 20% with maturation of all cell lines. The bone marrow contains less than 5% blast cells, and Auer rods is not detectable.
Time Frame: 7 days post completion of induction chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Idarubicin, Cytarabine)
Number analyzed (Participants) | 111
Participants
  CR | 77
  No CR | 32
  Unknown | 2

2. Secondary Outcome: Bone Marrow at Day 7 Post-Induction Chemotherapy
Description: Bone marrow positive, negative cells at day 7 post-induction chemotherapy for leukemia (%)
Time Frame: 7 days post completion of induction chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Idarubicin, Cytarabine)
Number analyzed (Participants) | 111
Participants
  Positive for Leukemia | 17
  Negative for Leukemia | 90
  Unknown | 4

ADVERSE EVENTS:
Arm/Group | Treatment (Idarubicin, Cytarabine)
Serious Adverse Events (participants affected / at risk) | 51/111
Other Adverse Events (participants affected / at risk) | 95/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Idarubicin, Cytarabine) (N=111)
Infection (Infections and infestations) | 4 (4)
Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Liver (Hepatobiliary disorders) | 1 (1)
Lung (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 20 (20)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 10 (10)
Edema/Anasarca (Investigations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Pleuritic Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Idarubicin, Cytarabine) (N=111)
Infection (Infections and infestations) | 56 (56)
Skin (Skin and subcutaneous tissue disorders) | 70 (70)
Mucositis (Gastrointestinal disorders) | 43 (43)
Renal (Renal and urinary disorders) | 22 (22)
Liver (Hepatobiliary disorders) | 59 (59)
Lung (Respiratory, thoracic and mediastinal disorders) | 32 (32)
Heart (Cardiac disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 75 (75)
Vomiting (Gastrointestinal disorders) | 66 (66)
Diarrhea (Gastrointestinal disorders) | 66 (66)
Fever (General disorders) | 66 (66)
Hemorrhage (Blood and lymphatic system disorders) | 15 (15)
Anxiety (Nervous system disorders) | 10 (10)
Headache (Nervous system disorders) | 24 (24)
Fatigue (General disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 9 (9)
Chills (General disorders) | 11 (11)
Edema (General disorders) | 8 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (7)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes